CLINICAL TRIAL: NCT03095586
Title: Interpretation of Health News Items Reporting Results of Randomized Controlled Trials With or Without Spin: A Randomized Controlled Trial Among English-speaking Patients
Brief Title: Interpretation of Health News Items Reporting Results of Randomized Controlled Trials With or Without Spin by English-speaking Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Isabelle BOUTRON, Professor, Assistance Publique - Hôpitaux de Paris
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ISB-009
Record Dates: First submitted 2017-03-24; First posted 2017-03-29 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: The Study Focus on no Specific Condition
Keywords: Spin; Misleading reporting; Misleading interpretation; Misleading extrapolation; Randomized controlled trials; Patients
MeSH Terms: interventions — spindlin

STUDY DESIGN:
Intervention Model Description: Two arms, parallel group, randomized controlled trial
Who Masked: Participant
Masking Description: Participants will be blinded to the study hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- News with Spin (Active Comparator): News items reporting results of RCTs with spin
  Interventions: Other: News items with spin
- News without spin (Experimental): News items reporting results of RCTs without spin
  Interventions: Other: News items without spin

INTERVENTIONS:
Other: News items with spin — Interpretation of news items with spin
  Arms: News with Spin
Other: News items without spin — Interpretation of news items without spin
  Arms: News without spin

SUMMARY:
The main objective of this study is to compare the interpretation of health news items reporting results of randomized controlled trials (RCTs) with or without spin (i.e., distortion of research results). The news items which reported those studies evaluating the treatment effect, having highest number of spin in the headline and text and received high online public attention will be selected. Spin will be deleted and will rewrite the news items without spin. This sample of news items reporting results of RCTs with and without spin will be interpreted by English-speaking patients.

DETAILED DESCRIPTION:
Health news is an important way to communicate updated medical research to the public. News items reporting the results of medical research attract a large audience. However, the quality of reporting in health news is questionable. The merits of a wide range of treatments and tests are overplayed and harms are underplayed. Several studies have shown the presence of spin (i.e., distorted presentation of study results) in health news. Distorted facts can be misleading and can affect the behaviour of physicians, healthcare providers and patients. However, little research has assessed whether spin can affect readers' interpretation of health news items.

Objective: "Spin" is defined as a misrepresentation of study results whatever the motive (intentionally or unintentionally) to highlight that the beneficial effect of the intervention in terms of efficacy and safety is greater than that shown by the results. To compare the interpretation of health news items reporting RCTs with or without spin. News items evaluating the effect of a pharmacological treatment that received high online public attention will be focused.

Hypothesis: The hypothesis of this study is that the spin can influence the reader's interpretation of health news items reporting results of RCTs.

Design: A randomized controlled trial

1. Interventions: Health news items reporting results of RCTs with and without spin will be compared. A sample of health news items reporting the results of RCTs evaluating the effect of pharmacologic treatment and containing highest number of spin in the headline and text will be selected. Spin will be deleted in the selected news items and will be rewritten the news items without spin.
2. Participants: The participants will include English-speaking patients from an online patient community.
3. Sample size: The sample size will be 300 patients.
4. The primary outcome will be perception of beneficial effect of the treatment X. We will ask participants, what do you think is the probability that treatment X would be beneficial to patients? (scale, 0 [very unlikely] to 10 [very likely]). Perception of safety and beneficial effects of treatment in clinical studies is considered as a surrogate marker of health outcome as it may have an impact on the future development of the drug, and then the potential use of the drug for patients.
5. Expected results: This study will evaluate the impact of spin on the interpretation of news items reporting results of RCTs by English-speaking patients.
6. This study is approved by ethics review regulations by INSERM (CEEI-IRB): IRB00003888

ELIGIBILITY:
Inclusion Criteria:

* Native English speakers or have a very good level in reading and understanding of English language
* Have at least one chronic disease

Exclusion Criteria:

-

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Perception of beneficial effect of the treatment X | As the intervention is assigned (reading the news item) i.e., 1-2 hours
  We will ask participants, what do you think is the probability that treatment X would be beneficial to patients? With the choices of answers on a 10 point Likert scale, (scale, 0 [very unlikely] to 10 [very likely])

SECONDARY OUTCOMES:
Perception of efficacy, safety, availability and clinical utility of the treatment X in existing clinical practice | As the intervention is assigned (reading the news item) i.e., 1-2 hours
  We will ask participants, what do you think is the size of the potential benefit for patients? With the choices of answers on a 5 point scale (scale, [none, small, moderate or large])
How safe do you think that treatment X would be for patients? | As the intervention is assigned (reading the news item) i.e., 1-2 hours
  With the choices of answers on a 10 point Likert scale, (scale, 0 [very unsafe] to 10 [very safe]) analysis: none, small vs moderate or large
Do you think this treatment should be offered to patients in the short term? | As the intervention is assigned (reading the news item) i.e., 1-2 hours
  With the choices of answers on a 10 point Likert scale, (scale, 0 [absolutely no] to 10 [absolutely yes])
Do you think this treatment will make a difference in the existing clinical practice? | As the intervention is assigned (reading the news item) i.e., 1-2 hours
  With the choices of answers on a 10 point Likert scale, (scale, 0 [absolutely no] to 10 [absolutely yes])

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle BOUTRON, Prof., Principal Investigator — INSERM U1153, University of Paris-Descartes; Romana HANEEF, PhD researcher, Principal Investigator — INSERM U1153, University of Paris-Descartes
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boutron I, Haneef R, Yavchitz A, Baron G, Novack J, Oransky I, Schwitzer G, Ravaud P. Three randomized controlled trials evaluating the impact of "spin" in health news stories reporting studies of pharmacologic treatments on patients'/caregivers' interpretation of treatment benefit. BMC Med. 2019 Jun 4;17(1):105. doi: 10.1186/s12916-019-1330-9. PMID 31159786